CLINICAL TRIAL: NCT03982082
Title: Feasibility Study of Ultrasound to Evaluate Muscle-Glycogen Content in Patients With Cancer
Brief Title: Ultrasound in Evaluating Muscle-Glycogen Content in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-1180; NCI-2019-02281 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1180 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-04-23; First posted 2019-06-11 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cachexia; Malignant Solid Neoplasm
MeSH Terms: conditions — Cachexia | interventions — Physical Therapy Modalities; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device feasibility (MuscleSound technology) (Experimental): Patients undergo ultrasound via MuscleSound technology over 3 minutes at baseline and immediately after each of 2 physical therapy sessions comprising cycling or walking over 10 minutes.
  Interventions: Procedure: Physical Therapy; Other: Questionnaire Administration; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Physical Therapy — Undergo physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Ultrasound — Undergo ultrasound via MuscleSound technology

SUMMARY:
This trial studies how well an ultrasound procedure (non-invasive MuscleSound technology) can be used to learn about levels of glycogen (a type of sugar) in cancer patients during inpatient rehabilitation. The ultrasound information will be processed to represent the energy storage in the muscle. The energy storage in the muscle may help future research to look for dietary plans that can help to increase energy storage, patient exercise tolerance, and functional improvement.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine feasibility of using non-invasive MuscleSound technology to determine glycogen stores in cancer patients.

EXPLORATORY OBJECTIVES:

I. Determine the baseline glycogen storage in two different groups of cancer patients, who are undergoing inpatient rehabilitation: (1) those with cachexia; (2) those without cachexia.

II. Determine the rate of depletion of muscle-glycogen stores by calculating the "Fuel Rating" score (FRS) at baseline, after 10-min of exercise and then again after 20-min of exercise.

III. Determine if there is any correlation between muscle-glycogen (at baseline and its depletion rate over time) and other factors including cancer type, cancer stage, patient age, patient sex, current body mass index (BMI), presence or absence of cachexia, functional measures and patient reported outcomes.

OUTLINE:

Patients undergo ultrasound via MuscleSound technology over 3 minutes at baseline and immediately after each of 2 physical therapy sessions comprising cycling or walking over 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to give written informed consent and to comply with study procedures.
* Patients with a biopsy-confirmed solid malignant neoplasm with at least one neurologically-intact lower extremity, who fit into one of the following groups:

  * Group 1: Patients with cachexia, defined by loss of > 5% of body weight over the preceding 6-months (in absence of simple starvation defined as intentional weight loss) or weight loss > 2% with BMI < 20.
  * Group 2: Patients without cachexia, as defined above.
* Patients who have a record of weight or BMI over preceding 6-months.
* Patients must be receiving rehabilitation that includes exercise under the direction of a physical therapist.

Exclusion Criteria:

* Non-English speaking patients.
* Patient with neurological compromise of both lower extremities causing muscle atrophy.
* Underlying unstable medical condition (i.e: cardiac, pulmonary, or hematological) or musculoskeletal injury, which in the opinion of the investigator, limits participation in exercise of the measured lower extremity.
* Patients who are unable to understand or follow through with study instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Glycogen Storage Assessment | Within 30 minutes of consent
  Muscle-glycogen status will be assessed using ultrasound and MuscleSound® technology which generates an average FRS (Fuel Rating Score)

OTHER OUTCOMES:
Functional Independent Measure | At baseline
  The FIM (Functional Independent Measure) score will be collected retrospectively from the patient's medical record as this is performed by a nurse or therapist. This measure provides a measurement for assessing how much assistance is required for the patient to complete activities of daily living.
Cancer characteristics of the patient | At baseline within 30 minutes of consent
  Type of cancer, stage of cancer; past and present treatment
Patient reported outcomes | At baseline
  Patient-Generated Subjective Global Assessment (PG SGA-SF) Patient Reported Outcomes is a tool used to measure risks for malnutrition.
Patient reported outcomes | At baseline
  Edmonton Symptom Assessment Scale (ESAS) is a validated tool for regular assessment of symptom distress in the Rehabilitation setting. Patients are asked to grade severity of their symptoms from "no symptom" 0 to "worst symptom" 10 in the last 24 hours. ESAS has high test-retest reliability of (>0.8) and has been validated in many clinical settings including cancer patients.
Body Composition | At baseline
  Will be accessed using the bioimpedance machine to measure body fat and muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Guo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03982082/ICF_000.pdf